## CLINICAL INSTRUMENTAL EVALUATION OF THE EFFICACY OF A COSMETIC PRODUCT IN IMPROVING SKIN MOISTURIZATION AND SKIN BARRIER

**Protocol ID:** IT0007726/24

**Date:** 15Dec2024

## **Study synopsis**

The study was aimed to assess the efficacy of a cosmetic product in improving skin moisturization and skin barrier function. In order to reach this goal a randomized, clinical trial was conducted on 30 (35 enrolled) healthy female and male subjects between 18 and 65 years old, enrolled according to the specific inclusion and non-inclusion criteria. The subjects had dry, very dry, sensitive and cracked skin showing discomforts related to this skin conditions (skin dryness, desquamation, skin tightness, and itching). According to a previously defined randomization list subjects applied tested product on right or left leg, and the other leg was left untreated and act as control area. The study duration was 28 days with evaluations performed at baseline (T0), after 30 minutes (T30min), 24 hours (T24h), 48 hours (T48h) from the first product application and after 7 (T7) and 28 days (T28) of product use. An independent ethics committee approved the study.